CLINICAL TRIAL: NCT07024979
Title: The Effects and Hyperscanning-Based Neural Mechanisms of Music Therapy on Social Relationships and Mental Wellness in University Students: A Randomized Controlled Trial
Brief Title: Music Therapy's Impact on University Students' Social and Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA240556
Record Dates: First submitted 2025-05-12; First posted 2025-06-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2024-12

CONDITIONS: Depressive Symptoms; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the intervention's inherent characteristics, complete blinding is not feasible for music therapists and investigators. The therapeutic nature of songwriting requires therapist awareness, while control condition procedures maintain equivalent therapist presence without therapeutic techniques. All analyses will be conducted with assessors maintain blinding until completion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy Songwriting Intervention (Experimental): This arm of participants will be receiving individual music therapy songwriting intervention as intervention.
  Interventions: Behavioral: Music Therapy Songwriting Intervention
- Non-therapeutic Music Listening and Discussion (No Intervention): This arm of participants will receive non-therapeutic music listening and discussion (non-therapeutic topics/techniques) sessions as the control condition. This active control condition matches the experimental intervention in format and include musical element, but excludes therapeutic components. The music therapist will ask the participant to provide 3 to 4 their preferred songs. Then they will listen to these songs through standardized equipment. Following each song, the therapist facilitates a structured discussion focused on normal domains and non-therapeutic topics, such as music styles, tempos, and factual information about artists and genres.

INTERVENTIONS:
Behavioral: Music Therapy Songwriting Intervention — The music therapy songwriting intervention is an active, client-centered music therapy approach in which the participant collaboratively create an original song with a professional music therapist. This evidence-based method combines: 1) lyric writing: the participant can express personal experience/emotions through guided lyric creation; 2) musical composition: the participant will choose or improvise their favorite melody, harmony, and rhythm with a music therapist; 3) therapeutic processing: discussion of song meaning and emotional connections between the participant and music therapist.
  Arms: Music Therapy Songwriting Intervention

SUMMARY:
In recent years, university education has become more challenging due to increased academic competition. A rising number of university students globally are currently being diagnosed with mental health problems, and previous research suggests that insufficient social support plays a significant role in the development of mental illnesses, such as symptoms of depression and anxiety. Music Therapy has been widely used in emotional regulation, offering a promising solution for people struggling with anxiety, depression, and social isolation. Research on the neural mechanisms underlying music therapy represents rapidly growing field of study. Hyperscanning is one of the useful neuroscience study methods, which is widely-used for study interbrain synchronization, refers to the simultaneous measurement of brain activity in two or more individuals who are interacting with each other. This study aims to investigate the effectiveness of music therapy intervention in enhancing mental health and social skills of university students with depressed, anxious, and stress symptoms. This current study will adopt a 2-arm randomized controlled design comparing therapeutic songwriting (experimental condition) with non-therapeutic music listening and discussion (control condition). Upon screening for inclusion criteria, baseline data will be collected; and eligible participants will be randomized into either 4 individual music therapy sessions or non-therapeutic music listening and discussion sessions.

DETAILED DESCRIPTION:
A rising number of university students globally are currently being diagnosed with mental health problems, and previous research suggests that insufficient social support plays a significant role in the development of mental illnesses, such as symptoms of depression and stress. Recent research indicates that 2.6% of young people worldwide experience depression, which is often associated with insufficient social interactions, challenges in emotional regulation, and unhealthy social relationships. These challenges may further impact their educational attainment, mental well-being, and quality of life. To address the impairment of mental health problems and its related influence on youths and their families, researchers, psychiatrists, and clinical therapists have been exploring innovative treatment approaches. Music therapy is one of these approaches.

In recent years, researchers have shifted their focus from simply demonstrating the effectiveness of music therapy treatment toward a deeper exploration of the underlying mechanisms of music used in these interventions. The field of research on Interbrain Synchronization (IBS) offers valuable insights into the intricate neural activities occurring across different brains and brain regions during human interaction. Hyperscanning, a widely-used method for studying interbrain synchronization, refers to the simultaneous measurement of brain activity in two or more individuals who are interacting with each other through various techniques, such as functional magnetic response imaging (fMRI), electroencephalography (EEG), magnetoencephalography (MEG), and functional near-infrared spectroscopy (fNIRS). The use of hyperscaning methods during clinical music therapy sessions may provide the opportunity to understand how music interventions affect the neural connections between therapist and client during a real clinical environment. However, a limited number of studies specifically examine this phenomenon within the unique setting of music therapy.

This study aims to bridge the gap between neuroscience, clinical music therapy, social relationships, and mental health by investigating the effects of EEG interbrain synchronization in undergraduate students. It seeks to explore further the connections between music, the brain, and psychological well-being, aiming to understand the underlying neurological mechanism.

This current study will adopt a 2-arm randomized controlled design comparing therapeutic songwriting (experimental condition) with non-therapeutic music listening and discussion (control condition). To address the research objectives, this study will track psychological and neurophysiological changes across four individual sessions through a combination of repeated measures. Participants and music therapists will wear synchronized EEG caps during each session to capture interbrain dynamics, while participants complete post-session therapeutic relationship and satisfaction ratings. Mental health outcomes will be assessed using standardized questionnaires administered at baseline (pre-intervention) and immediately following the final session (post-intervention). This multi-method approach integrates: 1) temporal tracking of psychological changes (both immediate session-level effects and cumulative intervention effects), 2) objective neurophysiological data on therapeutic rapport, and 3) subjective evaluations of the therapeutic process, collectively provide a multidimensional understanding of music therapy mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* (1) adults who aged between 18-40
* (2) without any mental diagnosis
* (3) able to speak and read Mandarin, Cantonese, or English
* (4) moderate stress or problems in academic activities, problems in interpersonal relationships, or adaptability to college life.
* (5) participants DASS-21 score >= "Moderate" severity on each subscale (Depression >= 14; Anxiety >= 10; Stress >= 19).

Exclusion Criteria:

* (1) has more than 10 consecutive years professional music training
* (2) with chronic illness and taking medication
* (3) with prior history of brain trauma or brain surgery
* (4) wearing metal piercings or implants.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Baseline Depression Anxiety Stress Level after 4 Sessions | Baseline (day 1), and the last session (up to 2 weeks, the 4th session)
  English and administration of the Chinese translated version of The Depression Anxiety and Stress Scale-21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content.
  The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest, anhedonia and inertia.
  The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect.
  The stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable/over-reactive and impatient.
  Scores of depression, anxiety, and stress are calculated by summing the scores for the relevant items.
Change of Baseline Social Connection Level after 4 Sessions | Baseline (day 1), and the last session (up to 2 weeks, the 4th session)
  English and administration of the Chinese translated version of the UCLA-Loneliness Scale (ULS-8).
  ULS-8 has been used to evaluated severity of feelings of loneliness in individuals, from adolescence to adulthood.
  Scale consists of 8 items which were loaded into a single factor. ULS-8 is a Likert-type scale with 4 options "(1) Never, (2) Rarely, (3) Sometimes and (4) Always". "I am an extrovert person" and " I can find friends when I want" items are reverse-scored.
  Sum of 8 items reveal general loneliness score, minimum and maximum possible scores are 8 and 32, respectively, higher scores from USL-8 correspond to severe loneliness in adolescents and young adults.
Interbrain Synchrony Level During 4 Sessions (EEG-based) | Baseline (day 1), the 2nd session (3 days after the first session), the 3rd session (at the beginning of the second week) , the 4th session (3 days after the 3rd session, up to two weeks).
  The interbrain synchronization level between the participant and music therapist in 4 sessions.
  EEG will be simultaneously recorded from both participants using two electrode caps with 16 Ag/AgCl electrode each. The electrode placement will follow the international 10-20 system guidelines.
  The EEG LAB toolbox and in-house scripts for MATLAB will be used for data processing. Specifically, phase locking value (PLV) and partial directed coherence (PDC)will be used to examine the magnitude of phase synchrony and its directionality, respectively during sessions. The connectivity analysis will be performed with the FieldTrip toolbox. The PLV quantified the degree of IBS between individuals.
Change of Baseline Hospital Anxiety and Depression Scale | Baseline (day 1), and the last session (up to 2 weeks, the 4th session)
  English and administration of the Chinese translated version of the Hospital Anxiety and Depression Scale (HAD-14) is a 14-item self-report questionnaire designed to screen for symptoms of anxiety and depression in non-psychiatric medical settings. It consists of two subscales (7 items measuring anxiety and 7 items measuring depression). Each item is rated on a 4-point scale (0 = not at all, 3 = nearly every day), with subscale scores ranging from 0 to 21 for each domain. Higher score indicates more severe symptoms.
Change of Baseline Perceived Stress Level | Baseline (day 1) and the last session (up to 2 weeks, the 4th session)
  English and administration of the Chinese translated version of the Perceived Stress Scale (PSS-10) will be used in this study. PSS-10 has been widely used to assess the degree to which individuals perceived their lives as unpredictable, uncontrollable, and overloaded in the past month. Comprising 10 items rated on a 5-point Liker scale (0 = never to 4 = very often). Total scores range from 0 to 40, with higher scores indicating higher levels of perceived stress.

SECONDARY OUTCOMES:
Work Alliance After Each Session | Baseline (day 1), the 2nd session (3 days after the first session), the 3rd session (at the beginning of the second week) , the 4th session (3 days after the 3rd session, up to two weeks).
  English and administration of the Chinese translated version of the Work Alliance Inventory-Short Revised (WAI-SR).
  The WAI-SR is a 12-item measure for the assessment of the therapeutic alliance. It assesses three key aspects of the therapeutic alliance (1) agreement on the tasks of therapy, (2) agreement on the goals of therapy and (3) development of an affective bond.
Therapeutic Rapport After Each Session | Baseline (day 1), the 2nd session (3 days after the first session), the 3rd session (at the beginning of the second week) , the 4th session (3 days after the 3rd session, up to two weeks).
  English and administration of the Chinese translated version of the Session Rating Scale (SRS).
  The SRS is a simple, 4-item visual analogue scale designed to assess key dimensions of effective therapeutic relationships.
  The SRS translates what is known about the alliance into four visual analogue scales each 10cm long to assess the clients' perceptions of: (1) respect and understanding, (2) relevance of the goals and topics, (3) client-practitioner fit and (4) overall alliance.
The Participant's State Anxiety After Each Session | It will be used to assess the participant's anxiety levels before and after each session, so the assessment will occur at the beginning and after each session, pre and post session 1, pre and post session 2, pre and post session 3, pre and post session 4
  The participant's state anxiety will be assessed after each session with the English and Chinese version of State-Trait Anxiety Inventory (STAI)-State Anxiety Subscale (Form Y-1). The STAI for Y-1 is a 20-item self-report measure designed to evaluate transient feelings of anxiety experience in the moment. Each item is rated on a 4-point Liker scale (1 = not at all to 4 = very much to), with statements reflecting current emotional states. Total scores range from 20 to 80, with higher scores indicating greater state anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Wanru Zhao, Principal Investigator — The University of Hong Kong
Locations (1):
- 2/F., The Hong Kong Jockey Club Building for Interdisciplinary Research, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
This study is committed to transparent and ethical data sharing to advance scientific collaboration while protecting participant confidentiality. The sharing data include assess to the study protocol, statistical analysis plan, and de-identified participant data.
  1. Full study protocol will be shared or published as a supplement to the primary trial manuscript in a public registry. It will available upon trial completion or concurrent with the first results publication.
  2. Primary and secondary outcome analyses data will be upload to journal supplementary materials. Finalize before database lock and shared with manuscript submission.
  3. De-identified participant data will be shared to researchers with reasonable requests, such as meta-analysis.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol will be shared upon trial completion or concurrent with the first results publication. The statistical analysis plan will be shared before database lock and shared with manuscript submission.
Access Criteria: Academic researchers affiliated with recognized institutions (universities, hospitals, NGOs) with reasonable requests.